CLINICAL TRIAL: NCT05939427
Title: Real-Time Feedback to Improve Family Engagement in Acute Cardiovascular Care
Brief Title: Improving Family Engagement in Acute Cardiovascular Care: The NGAGE Trial
Acronym: NGAGE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lady Davis Institute (Other)
Responsible Party: Principal Investigator, Michael Goldfarb, Clinician-Investigator, Lady Davis Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2023-3590
Record Dates: First submitted 2023-07-02; First posted 2023-07-11 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Family Engagement

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- NGAGE tool group (Experimental): Will have access to the NGAGE tool to learn about engaging in care and to request engagement activities.
  Interventions: Other: NGAGE tool
- Non-Intervention (No Intervention): Will receive usual care standards.

INTERVENTIONS:
Other: NGAGE tool — Will have access to the NGAGE tool to learn about engaging in care and to request engagement activities.
  Arms: NGAGE tool group

SUMMARY:
The objective of this study is to assess if the NGAGE real-time feedback tool improves family engagement in family members of people admitted to an acute cardiac care unit

The investigators will randomize 88 family members of people hospitalized in the acute cardiac ward in a 1:1 manner to either the NGAGE intervention or usual care. Family members will be eligible if the expected unit stay of their loved one is >48 hours and if they can communicate in English or French. A family member is considered anyone with a biological, emotional, or legal relationship with the patient whom the patient wishes to be involved in their care. The primary outcome of the study will be the FAMily Engagement (FAME) score at hospital discharge. Secondary outcomes will be family mental health (by HADS score) and family care satisfaction (by FS-ICU score).

ELIGIBILITY:
Inclusion Criteria:

* Family member of CV patient with expected stay > 48 hours (as per treating team)
* Aged of at least 18 years old
* Ability to communicate in English or French
* Willing to fill out the questionnaires as per the study

Exclusion Criteria:

* Expected stay of < 48 hours
* Inability to communicate in English or French

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Family Engagement (FAME) score | Within 48-hours of hospital discharge
  An engagement score that measures the following domains: family presence, family needs, communication and education, decision making, and direct care. Family-centered care principles are also captured such as dignity and respect, information sharing, participation and collaboration. The score is continuous and ranges from 0 to 100, with higher scores indicating increased levels of care engagement.

SECONDARY OUTCOMES:
Mental health | Within 48-hours of hospital discharge
  The Hospital Anxiety and Depression Scale (HADS) is a self-reported tool to measure anxiety and depression. Scores range from 0-14 with higher scores indicating increased levels of anxiety and depression.
Family satisfaction | Within 48-hours of hospital discharge
  The Family Satisfaction in the Intensive Care Unit (FS-ICU) tool is used to assess the family satisfaction and experience with care in the ICU. Scores range from 0-100 with higher scores indicating increased family satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Goldfarb, MD, MSc, Principal Investigator — Lady Davis Institute, McGill University, Jewish General Hospital
Locations (1):
- Ladis Davis Institute, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No